CLINICAL TRIAL: NCT05545540
Title: Feasibility Study on the Antiseizure and Neurocognitive Effects of Musical Neurostimulation in Paediatric Patients With Drug Resistant Epilepsy
Brief Title: Music as an Adjunctive Epileptic Seizure Treatment Option
Acronym: MAESTRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1-106-22
Record Dates: First submitted 2022-09-14; First posted 2022-09-19 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Epilepsy; Neurocognitive Disorders
MeSH Terms: conditions — Epilepsy; Neurocognitive Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Patients will be issued Mp3 players and speakers with music files in Mp3 formatted by the randomization team. The intervention arm will be issued the first movement (8 minutes, 22 seconds) of Mozart's Sonata for Two Pianos in D Major, K448. They will be exposed to it once a day during wakefulness for two consecutive months.
  Interventions: Other: Musical Neurostimulation
- Control arm (Placebo Comparator): Patients will be issued Mp3 players and speakers with music files in Mp3 formatted by the randomization team. The control arm will receive the first movement (8 minutes, 34 seconds) of Mozart's Fantasia for Piano in C Minor, K 475. Although from the same composer, the control sonata has been found not to have neurostimulating properties. They will be exposed to it once a day during wakefulness for two consecutive months.
  Interventions: Other: Placebo Musical Neurostimuloation

INTERVENTIONS:
Other: Musical Neurostimulation — Daily exposure to musical composition found to have antiseizure properties
  Arms: Intervention arm
Other: Placebo Musical Neurostimuloation — Daily exposure to musical composition found NOT to have antiseizure properties
  Arms: Control arm

SUMMARY:
Mozart's Sonata for two pianos in D major (K448) has been found to reduce the presence of abnormalities in the electroencephalograms of patients with epilepsy. We will examine the long term effects of listening to the K448 sonata on seizure frequency and cognitive functioning in children with drug resistant epilepsy allocated to either a study group or a control group. Patients' parents will complete a seizure diary for the whole study period, during which antiepileptic drug therapy of the child will remain unchanged. Baseline neuropsychological testing will be performed and a seizure diary will be kept for 3 months. The study group will listen to K448 for 8 continuous minutes every day for 2 months, while those in the control group will listen to control music for the same amount of time. Neuropsychological testing will be repeated at the end of the study period and any change from baseline examined. Seizure frequency during periods of exposure to music will be compared to baseline in both groups. Feedback questionnaires and parent focus groups will be used to gather information around the practicalities of exposure to music, potential problems and suggestions for how future studies might be improved.

DETAILED DESCRIPTION:
Primary Objectives:

(i) Determine feasibility of a double-blind, randomized, study on the epileptological and neuropsychological effects of Mozart's K448 sonata on paediatric drug resistant epilepsy (ii) Ascertain the logistical and methodological challenges that need to be addressed in order for a definitive study to be designed and conducted (iii) Determine what recruitment criteria and patient numbers are necessary to ensure such a fully powered study

Primary Outcome:

The primary outcome measure is seizure frequency after exposure to Mozart's K448 sonata.

Secondary Outcome:

Initial and re-test scores on age-appropriate tests of cognitive functioning, and initial and re-test scores on measures of adaptive behaviour and quality of life.

Study Description Patient demographic and clinical data will be recorded prior to study onset and parents will be issued diaries to record seizures and music exposure (date, time of day, duration) during the intervention phase. Parents will be asked to fill out diaries for one month prior to music exposure, for the two-month musical intervention period and one month after the intervention period.

Patients will be randomly allocated 1:1 to either the intervention or the control arm by using a remote central computer-generated randomisation schedule hosted at the University of Aberdeen Clinical Trials Unit (CHaRT). Parents will be issued Mp3 players and speakers with music files in Mp3 formatted by CHaRT. The intervention arm will be issued the first movement (8 minutes, 22 seconds) of Mozart's Sonata for Two Pianos in D Major, K448. The control arm will receive the first movement (8 minutes, 34 seconds) of Mozart's Fantasia for Piano in C Minor, K 475. Although from the same composer, the control sonata has been found not to have neurostimulating properties.

Parents will be asked to play the assigned music to their child while awake once a day, every day, for two consecutive months. Freedom will be given regarding time of day, as long as the child is awake and is not exposed to interfering noise or music. Parents will be told to keep the speakers at a minimum distance of 1 meter from the child, with a volume setting corresponding to 75 dB.

Seizure data Diaries will record seizure data for one month before the musical intervention, two months during intervention and for one month after the intervention. This will include date and time of onset, duration and seizure type.

Caring clinicians will be asked to annotate clinical events that might have had an impact on seizure threshold during the study period on appropriate data request forms.

Neuropsychological functioning All children will have their cognitive functioning assessed at baseline and at the end of the intervention period (i.e. two months later). For children aged 2 to 2½ years, specific subtests from the Bayley Scales of Infant and Toddler Development-Third Edition, Screening Test (Bayley-III Screening Test) will be administered. For children aged between 2½ and 7½ years, specific subtests from the Wechsler Preschool & Primary Scale of Intelligence-Fourth Edition (WPPSI-IV) will be administered, while children aged over 7½ years will receive specific subtests from the Wechsler Intelligence Scale for Children-Fifth Edition (WISC-V).

The Bayley-III Screening Test (Bayley, 2006) is an individually administered instrument designed to briefly assess the cognitive, language and motor functioning of infants and young children between 1 month and 42 months of age. Individual subtests evaluate aspects of Cognitive development (33 items), Receptive Communication (24 items), Expressive Communication (24 items), Fine Motor skills (27 items), and Gross Motor skills (28 items). The primary purposes are to determine quickly whether a child is progressing to normal expectations and to determine if more comprehensive evaluation is needed. The Cognitive, Receptive Communication, and Expressive Communication subtests will form key outcome variables for this study.

The WPPSI-IV (Wechsler, 2012) is an individually administered clinical instrument for assessing the cognitive abilities of children aged between 2 years 6 months and 7 years 7 months. It consists of a broad range of verbal and nonverbal/perceptual-motor subtests that contribute to the production of five primary index scores that represent intellectual functioning in specified cognitive domains (i.e. the areas of Verbal Comprehension, Visual Spatial functioning, Fluid Reasoning, Working Memory, and Processing Speed). The sum of an individual's performance across four subtests is used to calculate an additional composite (or index) score that represents a child's general intellectual ability (termed the GAI: General Ability Index). Four subtests require to be administered in order to obtain the GAI (a key outcome variable for this study).

The WISC-V (Wechsler, 2014) is an individually administered, comprehensive clinical instrument for assessing the intelligence of children aged between 6 years 0 months and 16 years 11 months. It is a comprehensive instrument in that it consists of a broad range of verbal and perceptual-motor subtests that contribute to the production of four composite or index scores that represent intellectual functioning in specified cognitive domains: Verbal Comprehension (VCI), Perceptual Reasoning (PRI), Working Memory (WMI), and Processing Speed (PSI). The sum of an individual's performance across these domains is used to calculate an additional composite (or index) score that represents a child's general intellectual ability. This is termed the General Ability IQ (GAI). Five subtests require to be administered in order to obtain the GAI (a key outcome variable for this study).

All test measures are well standardised clinical tools. In total, the time commitment required from child participants should be no longer than 30-35 minutes (on each occasion).

In addition to the above, parents will be asked to complete three questionnaires - at baseline and at the end of the intervention period - as an additional means to quantifying the potential impact of treatment on the child's psychosocial functioning/ wellbeing and adaptive behaviour:

1. Paediatric Quality of Life Inventory Epilepsy Module (PedsQL-Epilepsy Module) is a disease-specific health-related quality of life (QoL) measure designed to be used with children and young people with epilepsy. Using a 5-point Likert-scale, the 22 to 29-item parent-report version used for the purpose of this study evaluates the extent to which epilepsy and/or its treatments affect a child/ young person's QoL, with five key domain scores produced: this covering Mood/Behavioural functioning; Sleep/Fatigue; Executive Functioning; Cognitive functioning; and broader psychosocial Impact. Normative data is used for the purpose of comparison and determining the degree of abnormal functioning within each domain. This questionnaire takes no longer than 5 minutes to complete.
2. The Behavior Rating Inventory of Executive Function - Second Edition (BRIEF-2) is an established, reliable, and well-validated rating scale that evaluates a range of everyday behaviours that are associated with particular executive functioning abilities, including (i) inhibition, (ii) self-monitoring, (iii) mental shifting, (iv) emotional control, (v) initiation, (vi) working memory, (vii) planning, (viii) task-monitoring, and (ix) organisation of materials. It is designed to be used to provide commentary on a broad range of children for whom there may be concerns about self-regulation. The 63-item parent report version of the scale is to be used as part of the current study. This questionnaire takes no longer than 5 minutes to complete.
3. Adaptive Behaviour Assessment System - 3rd Edition (ABAS-3; Harrison & Oakland, 2015). The ABAS-3 provides a complete assessment of adaptive skills across the life span (from birth to 89 years). For children and young people, behaviour ratings are completed by a parent/ caregiver and/or a teacher; there is no self-report option for children and young people. For the 10 skill areas assessed (Communication, Community Use, Functional Academics, Home Living, Health and Safety, Leisure, Self-Care, Self-Direction, Social, and Work), norm-referenced scaled scores and test score age-equivalents can be derived. Scores in particular skill areas contribute to the calculation of three Adaptive Domain scores (Conceptual, Social, and Practical), while a General Adaptive Composite (GAC) score - that is based upon the sum of scores from 9 of the 10 core skill areas (i.e. excluding Work) - can also be calculated. This questionnaire should take no longer than 20 minutes to complete.

All assessments will be administered by a suitably qualified Research Assistant and completed by those children that participate in the study in an appropriate location; such as a quiet room at their school or a private consulting room at a convenient medical facility (such as their local health centre or treating hospital). Complete privacy will be required during this process. Child participants will be assessed on all measures twice; with an approximate 2 month gap between initial testing and follow-up testing. In total, the time commitment required from child participants should be no longer than 30-35 minutes (on each occasion). In line with this, parents should take no longer than 30-35 minutes to complete the required questionnaires (on each occasion).

Parental feedback Three groups of 8-10 participating parents will be invited to participate in focus interviews to provide their in-depth opinions and experiences on the pre-intervention, during intervention and post intervention phases. Topics covered will include compliance and reactions of their child with exposure to music, use of the equipment (eg. Mp3 players), diary completion and expectations of the project. Questions on strengths of the study, potential difficulties with the protocol and any improvements will be included.

Themes identified during focus groups will be used to adjust the current protocol in future fully powered studies.

Qualitative analysis Qualitative data will be analysed using a simple thematic, narrative summary approach. Barriers and facilitators to the study design and implementation of the intervention will be grouped into key themes and summarised.

Data processing At randomisation, all participants will be given a unique study ID which will be used to link clinical and demographic data. Identifiable data will be kept in a locked filing cabinet on NHSG premises and only available to members of the research team. Analysis will be on anonymised data.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with drug resistant epilepsy as per International League Against Epilepsy criteria: failure of adequate trials of two tolerated and appropriately chosen and used anti-seizure medication (ASM) schedules to achieve sustained seizure freedom.

Exclusion Criteria:

* Children who undergo changes in ASM treatment during the study period.
* Children with a seizure frequency of less than two episodes per month.
* Children who underwent changes in ASM therapy less than one month before the study period.
* Children included in other clinical intervention studies at the time of recruitment.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-01-02 (Estimated); Study Completion 2024-02-02 (Estimated)

PRIMARY OUTCOMES:
Seizure Frequency | 4 months after recruitment
  Changes in epileptic seizure frequency before and after exposure to musical neurostimulation.

SECONDARY OUTCOMES:
Changes in cognitive functioning from baseline to follow-up (at 2 months) on the Bayley Scales of Infant and Toddler Development-Third Edition, Screening Test. | 4 months after recruitment
  The Bayley-III Screening Test (Bayley, 2006) is an individually administered instrument designed to briefly assess the cognitive, language and motor functioning of infants and young children between 1 month and 42 months of age. Scores range from 0 to 33 with higher scores descriptive of higher levels of competency in the skill being assessed. The Cognitive, Receptive Communication, and Expressive Communication subtests will form key outcome variables for this study.
Changes in cognitive functioning from baseline to follow-up (at 2 months) on the Wechsler Preschool & Primary Scale of Intelligence-Fourth Edition (WPPSI-IV). | 4 months after recruitment
  The WPPSI-IV is an individually administered clinical instrument for assessing the cognitive abilities of children aged between 2 years 6 months and 7 years 7 months. Scores are expressed as scaled scores (from 1 to 19) with higher scores representative of higher functioning in the domain being assessed. Six subtests from the WPPSI-IV will be administered to participants, with measures of visual working memory, processing speed, and general intellectual functioning being key outcome variables for this study.
Changes in cognitive functioning from baseline to follow-up (at 2 months) on the Wechsler Intelligence Scale for Children-Fifth Edition (WISC-V). | 4 months after recruitment
  The WISC-IV is an individually administered clinical instrument for assessing the intelligence of children aged between 6 years 0 months and 16 years 11 months. Scores are expressed as scaled scores (from 1 to 19) with higher scores representative of higher functioning in the domain being assessed. Seven subtests from the WISC-V will be administered to participants, with measures of visual working memory, processing speed, and general intellectual functioning being key outcome variables for this study.
Changes in cognitive functioning from baseline to follow-up (at 2 months) on the NEPSY-II. | 4 months after recruitment
  The NEPSY-II assess neuropsychological development in children aged 3 to 16 years. Scores are expressed as scaled scores (from 1 to 19) with higher scores representative of higher functioning in the domain being assessed. All participants over the age of 3 years will complete the Speeded Naming subtest from the NEPSY-II, which is a measure of processing speed.
Changes in cognitive functioning from baseline to follow-up (at 2 months) on the Test of Everyday attention for Children (TEA-Ch). | 4 months after recruitment
  The TEA-Ch is a clinical battery of tests for children aged between 6 years and 16 years that allows for relative assessment across different attentional capacities. Scores are expressed as scaled scores (from 1 to 19) with higher scores representative of higher functioning in the domain being assessed. All participants over the age of 6 years will complete the Score! subtest from the TEA-Ch, which is a measure of sustained auditory attention.
Changes in psychosocial functioning from baseline to follow-up (at 2 months) on measures of adaptive behaviour and quality of life. | 4 months after recruitment
  Parents will be asked to complete three questionnaires - at baseline and at the end of the intervention period - as an additional means to quantifying the potential impact of treatment on the child's psychosocial functioning/ wellbeing and adaptive behaviour. Measures to be used are well-validated clinical instruments that evaluate quality of life (Paediatric Quality of Life Inventory Epilepsy Module: PedsQL-Epilepsy Module), attention and conduct problems (Conners' Rating Scale-Revised: CRS-R) and adaptive behaviour (Adaptive Behaviour Assessment System - 3rd Edition: ABAS-3). Raw score change on each of these measures will form key outcome variables; with higher scores representing better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Domenico Serino, MD, Principal Investigator — University of Aberdeen, NHS Grampian
Locations (1):
- Royal Aberdeen Children's Hospital, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hughes JR. The Mozart Effect. Epilepsy Behav. 2001 Oct;2(5):396-417. doi: 10.1006/ebeh.2001.0250. PMID 12609277
- [Background] Leng X, Shaw GL, Wright EL. Coding of musical structure and trion model of cortex. Music Percept 1990;8(1):9-62.
- [Background] Leng X, McGrann JV, Shaw GL. Reversal of epileptic state by patterned electrical stimulation suggested by trion model calculations. Neurol Res. 1992 Mar;14(1):57-61. doi: 10.1080/01616412.1992.11740012. PMID 1351261
- [Background] Grylls E, Kinsky M, Baggott A, Wabnitz C, McLellan A. Study of the Mozart effect in children with epileptic electroencephalograms. Seizure. 2018 Jul;59:77-81. doi: 10.1016/j.seizure.2018.05.006. Epub 2018 May 9. PMID 29763803
- [Background] Lin LC, Lee WT, Wang CH, Chen HL, Wu HC, Tsai CL, Wei RC, Mok HK, Weng CF, Lee MW, Yang RC. Mozart K.448 acts as a potential add-on therapy in children with refractory epilepsy. Epilepsy Behav. 2011 Mar;20(3):490-3. doi: 10.1016/j.yebeh.2010.12.044. Epub 2011 Feb 2. PMID 21292560
- [Background] Sesso G, Sicca F. Safe and sound: Meta-analyzing the Mozart effect on epilepsy. Clin Neurophysiol. 2020 Jul;131(7):1610-1620. doi: 10.1016/j.clinph.2020.03.039. Epub 2020 Apr 30. PMID 32449680